CLINICAL TRIAL: NCT00093236
Title: Systemic Endothelial Consequences of Periodontal Disease
Brief Title: Impact of Gum Infection on Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23262; R01DE015345 (NIH)
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease; Periodontal Disease
MeSH Terms: conditions — Cardiovascular Diseases; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Periodontal Treatment (Experimental): Subjects will receive scaling, root planing and if needed periodontal surgery
  Interventions: Procedure: Early Periodontal Treatment
- Usual Dental Hygiene (Active Comparator): Subjects will receive routine oral hygiene
  Interventions: Procedure: Usual Dental Hygiene

INTERVENTIONS:
Procedure: Early Periodontal Treatment — Subjects will receive scaling and root planing at baseline. Three weeks after initiation of the study, they will return and be re-evaluated for the need for periodontal surgery. If indicated, they will then receive definitive periodontal surgery over the next 4 weeks. At the 12-week time point, periodontal surgery will be reevaluated and further therapy provided as needed and make repeated visits as needed to achieve periodontal health.comprehensive periodontal treatment
  Arms: Early Periodontal Treatment
Procedure: Usual Dental Hygiene — Subjects will receive routine oral hygiene visits at the 3 and 12-week time points. After a 12-week period (24 week time point) to allow healing and resolution of a systemic inflammatory state, patients will return for follow-up measurements of periodontal parameters, vascular function and inflammation.
  Arms: Usual Dental Hygiene

SUMMARY:
The purpose of this study is to determine the effect of gum infection on parameters of cardio-vascular disease.

DETAILED DESCRIPTION:
Epidemiological studies indicate that individuals with severe periodontal disease have significantly increased risk for cardiovascular disease. Periodontal disease, a chronic bacterial infection of the gums, is associated with recurrent bacteremia and a state of systemic inflammation that may convert endothelial cells to a pro-atherogenic phenotype with increased expression of inflammatory factors and loss of the anti-thrombotic, growth inhibitory, and vasodilator properties of the endothelium, including a decrease in the biological activity of nitric oxide. In human subjects, endothelial dysfunction has evolved into a well-accepted indicator of early atherosclerosis and predictor of increased cardiovascular disease risk. We have recently demonstrated a strong association between severe periodontal disease and endothelial vasomotor dysfunction in a case control study of otherwise healthy human subjects. In that study, periodontal disease was also associated with higher plasma levels of the acute phase reactant C-reactive protein (CRP). These results support the hypothesis that severe periodontal disease induces a state of systemic inflammation that impairs endothelial function, however, the cross-sectional design leaves open the possibility that confounding factors explain the results. We now propose to determine whether effective treatment of periodontal disease improves endothelial function (Aim 1) and reduces inflammation (Aim 2) in a randomized intervention study. Patients will receive comprehensive periodontal treatment designed to produce a state of periodontal health (scaling and root planing and periodontal surgery with re-treatment as needed) or routine oral hygiene and will be followed for 24 weeks. The study will examine endothelium-dependent brachial artery flow-mediated dilation, systemic markers of inflammation and endothelial activation (CRP, IL-6, myeloperoxidase, and ICAM-1), and oral markers of periodontitis (PGE2, myeloperoxidase, and pathogen DNA) before and after treatment. Compared to oral hygiene (which will stabilize, but not reverse periodontal disease), we hypothesize that comprehensive treatment of periodontal disease will improve endothelium-dependent dilation and reduce local and systemic inflammation. Further, we suggest that the degree of improvement in endothelial function will relate to the degree of reduction in specific markers of inflammation. Such results would provide much stronger evidence for causal links between periodontal disease, systemic inflammation, and endothelial dysfunction, a recognized surrogate for cardiovascular risk. The proposed studies will provide new insights into how periodontal disease contributes to cardiovascular disease risk in human subjects and may lead to new approaches to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The study seeks to enroll patients with periodontal disease and no other major co-morbidities including cardiovascular disease or other major medical problems.
2. In this intervention study, cigarette smokers will be permitted as justified below and randomized in stratified fashion to ensure equal numbers in the two treatment groups.

Exclusion Criteria:

1. Known cardiovascular disease including coronary heart disease, cerebral vascular disease, peripheral vascular disease, valvular heart disease, and congestive heart failure.
2. Major coronary risk factors including diabetes mellitus, hypertension, hypercholesterolemia requiring treatment according to the ATP-III guidelines.
3. Other major illness including cancer, liver disease, renal disease, pulmonary disease, chronic infectious disease (including HIV and hepatitis C infection), rheumatological disease, hematological disease, or any condition requiring hospitalization or chronic medical therapy.
4. Use of antibiotics within three months.
5. Use of oral contraceptives or hormone replacement therapy.
6. Major psychiatric illness requiring treatment or that might interfere with the ability to understand and cooperate with the protocol.
7. Ongoing drug or alcohol abuse.
8. Use of sildenafil (Viagra) within 7 days because of the risk of marked hypotension with nitroglycerin administration.
9. History of migraine headaches that might be exacerbated by nitroglycerin.
10. Use of cholesterol lowering therapy, angiotensin converting enzyme inhibitors (subjects should not be taking these drugs because they will have no history of cardiovascular disease risk factors).
11. Antioxidant vitamins (vitamin C or vitamin E) in doses exceeding the Recommended Dietary Allowances (RDA), (60 mg/day and 30 IU/day, respectively).
12. Pregnancy, as diagnosed by serum beta-hCG.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-09; Primary Completion 2011-04 (Actual); Study Completion 2012-12-08 (Actual)

PRIMARY OUTCOMES:
Periodontal disease progression | 3 wks, 12 wks, and 24 weeks
  Three weeks after initiation of the study, they will return and be re-evaluated for the need for periodontal surgery. If indicated, they will then receive definitive periodontal surgery over the next 4 weeks. At the 12-week time point, periodontal surgery will be reevaluated and further therapy provided as needed and make repeated visits as needed to achieve periodontal health. During this period, the Usual Hygiene Group will return for oral hygiene visits at the 3 and 12-week time points. After a 12-week period (24 week time point) to allow healing and resolution of a systemic inflammatory state, patients will return for follow-up measurements of periodontal parameters, vascular function and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Salomon Amar, DMD, Ph.D, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No